CLINICAL TRIAL: NCT02621749
Title: Cerebral Microembolism in the Critically Ill With Acute Kidney Injury: A Prospective Multi-Center Randomized Controlled Trial Comparing Continuous With Intermittent Renal Replacement Therapy.
Brief Title: Cerebral Microembolism in the Critically Ill With Acute Kidney Injury
Acronym: COMET-AKI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 199/2015
Record Dates: First submitted 2015-11-20; First posted 2015-12-03 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Embolism
MeSH Terms: conditions — Intracranial Embolism | interventions — Renal Replacement Therapy; Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRRT group (Active Comparator): the CRRT group receives continuous renal replacement therapy for acute kidney injury
  Interventions: Device: Renal replacement therapy
- IRRT group (Active Comparator): the IRRT group receives intermittent renal replacement therapy after termination of CRRT.
  Interventions: Device: Renal replacement therapy

INTERVENTIONS:
Device: Renal replacement therapy — Patients receive renal replacement therapy according to institutional standards
  Other Names: Hemodialysis

SUMMARY:
The primary objective of this study is to investigate the impact of continuous renal replacement therapy and intermittent renal replacement therapy on microbubble / cerebral microemboli generation in a cohort of critically ill patients with dialysis-dependent acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yrs.
* Signed IC

Exclusion Criteria:

* Heart disease (PFO, ASD, VSD, severe valvular disease)
* Atrial fibrillation
* Cerebrovascular pathology
* Missing temporal bone window
* Allergy to plastic contained in the investigative device (transcranial Doppler)
* Chronic kidney disease
* Pregnancy
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01; Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Cerebral Microembolic Load detected by Transcranial Doppler Ultrasound | During hemodialysis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Erdoes, MD, Principal Investigator — University of Berne
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Erdoes G, Uehlinger DE, Kobel B, Stucki MP, Wiest R, Stueber F, Fankhauser N, Jakob SM, Schefold JC. Cerebral microembolism in the critically ill with acute kidney injury (COMET-AKI trial): study protocol for a randomized controlled clinical trial. Trials. 2018 Mar 21;19(1):189. doi: 10.1186/s13063-018-2561-3. PMID 29562937